CLINICAL TRIAL: NCT02786251
Title: The Role of Brown Adipose Tissue in Triglyceride Clearance in People
Acronym: BAT-TG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201602059
Record Dates: First submitted 2016-05-20; First posted 2016-05-30 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT+ (Other): Individuals with significant amounts of BAT (>20 ml)
  Interventions: Other: Cold exposure; Other: Exposure to thermoneutral conditions
- BAT- (Other): Individuals with no/minimal amounts of BAT (<20 ml)
  Interventions: Other: Cold exposure; Other: Exposure to thermoneutral conditions

INTERVENTIONS:
Other: Cold exposure — During cold exposure intervention, we will use an individualized cold exposure protocol above the individual shivering threshold of each participant using liquid condition garments and a temperature controlled room.
Other: Exposure to thermoneutral conditions — For the thermoneutral conditions intervention, subjects will be exposed to thermoneutral conditions (~26-28°C).

SUMMARY:
The recent discovery of functional brown adipose tissue (BAT) in humans has led to a paradigm shift in adipose tissue biology; it is now believed that adipocytes may play a significant role in regulating substrate metabolism. Given that the resurgence in the interest in human BAT is still in its infancy, a number of fundamental questions pertaining to the role of BAT in human physiology remain unanswered. One area of particular importance, but poorly understood, is the potential effect of BAT on triglyceride (TG) metabolism. Data from a series of studies have found that BAT is inversely associated with adiposity, high blood lipids, and fatty liver in people. However, the role of BAT in the regulation of TG metabolism in people is not known. The overall goal of this study is to determine the physiological importance of the human BAT in TG metabolism. To this end, we are planning to study overweight/obese women with high amounts of BAT (BAT+, n=14) and with no/minimal BAT (BAT-, n=14) both under thermoneutrality and mild cold exposure (~2 weeks apart). The investigators hypothesize that BAT+ participants will demonstrate greater plasma very low-density lipoprotein triglycerides (VLDL-TG) clearance rate compared to BAT- participants, and higher expression of genes involved in lipid metabolism only in BAT (but not muscle and white adipose tissue). Infusion of stable isotope tracers and metabolic modeling techniques will be used to assess VLDL-TG kinetics. Positron emission tomography computed tomography will be used for the identification and quantification of BAT. Supraclavicular BAT, abdominal white adipose tissue, and skeletal muscle tissue biopsies during cold exposure and thermoneutral conditions in conjunction with molecular biology techniques will used to measure expression of genes involved in lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 and ≤65 years
* BMI 25.0-35.0 kg/m²

Exclusion Criteria:

* Men
* Previous bariatric surgery or gastrointestinal surgery
* Structured exercise >2 days/week for ≥35 min of intense exercise (e.g., jogging, activity that causes heavy breathing and sweating) or ≥150 min per week of moderate intensity exercise (e.g., brisk walking)
* Unstable weight (>5% change during the last 2 months before entering the study)
* Significant organ system dysfunction (e.g., diabetes requiring medications, severe pulmonary, disorders of the gastrointestinal tract, kidney or cardiovascular disease)
* Current cancer or cancer that has been in remission for <5 years
* Conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* Use of medications that are judged by the investigators to affect the study outcome measures or increase the risk of study procedures (e.g., anticoagulants) and that cannot be temporarily discontinued for this study
* Smoke cigarettes or use of illegal drugs
* Consumption of >14 units of alcohol (e.g., glass of wine or bottle of beer) per week
* Pregnant or lactating
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Rate of VLDL-TG clearance | 12 hours
  The rate of VLDL-TG clearance from plasma will be assessed using infusion of stable isotopes.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chondronikola, PhD, RDN, Principal Investigator — University of California, Davis
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chondronikola M, Yoshino J, Ramaswamy R, Giardina JD, Laforest R, Wahl RL, Patterson BW, Mittendorfer B, Klein S. Very-low-density lipoprotein triglyceride and free fatty acid plasma kinetics in women with high or low brown adipose tissue volume and overweight/obesity. Cell Rep Med. 2024 Jan 16;5(1):101370. doi: 10.1016/j.xcrm.2023.101370. PMID 38232692